CLINICAL TRIAL: NCT02660645
Title: Blue Light Cystoscopy With Cysview® Registry
Acronym: BLCCR
Status: Recruiting | Type: Observational
Sponsor: Photocure (Industry)
Collaborators: Catalyst Pharmaceutical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: BLCCR-001
Record Dates: First submitted 2016-01-06; First posted 2016-01-21 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer
Keywords: Cysview; Hexaminolevulinate; Hexvix; NMIBC; BLCC; Blue Light Cystoscopy with Cysview; Cystoscopy; TURBT; TUR; Fluorescent cystoscopy; Non-muscle invasive bladder cancer (NMIBC); Transurethral resection (TUR)
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — 5-aminolevulinic acid hexyl ester; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blue Light Cystoscopy with Cysview®: Bladder cancer patients who have undergone Blue light cystoscopy with Hexaminolevulinate hydrochloride (Cysview®) 100mg in 50 milliliters (mL) reconstituted solution instilled intravesically into bladder prior to cystoscopy in operating room (OR). Retention time: 1-3 hours. The Karl Storz D-Light C Photodynamic Diagnostic (PDD) system is used for the cystoscopy procedure at the OR examination.
  Interventions: Drug: Hexaminolevulinate hydrochloride (HCL); Device: Karl Storz D-Light C Photodynamic Diagnostic (PDD) system

INTERVENTIONS:
Drug: Hexaminolevulinate hydrochloride (HCL) — Instillation in bladder
  Other Names: Cysview®; Hexvix®
Device: Karl Storz D-Light C Photodynamic Diagnostic (PDD) system — Cystoscopy procedure

SUMMARY:
Registry study to gather more information on the current use of Blue Light Cystoscopy with Cysview (BLCC) in urologists' practices.

DETAILED DESCRIPTION:
Data will be captured on specific patient types undergoing Blue Light Cystoscopy with Cysview for known or suspected non-muscle invasive bladder cancer. Specific clinical questions will be asked.

1. What is the incremental detection rate with Blue Light Cystoscopy with Cysview over conventional white light cystoscopy in each of the seven (7) patient populations? Does this translate into lower recurrence/progression rate?
2. How do the six (6) tumor variables used in the European Association of Urology (EAU) risk tables (primary/secondary, recurrence rate, size, multifocality, grade, and history of carcinoma in situ (CIS))6 affect this incremental rate?
3. How does an abnormal cytology or positive or negative fluorescent in situ hybridization (FISH) affect the likelihood that Blue Light Cystoscopy with Cysview will detect more cancers than white light?
4. What are the performance characteristics of Blue Light Cystoscopy with Cysview within eight (8) weeks of Bacillus Calmette-Guérin (BCG) with respect to improved tumor detection and false positive rate compared to conventional white light cystoscopy?
5. What is the incremental Blue Light Cystoscopy with Cysview detection rate over random bladder biopsies alone in patients being evaluated for routine three month restaging (group 4) or occult disease (group 5)?
6. What are the performance characteristics of Blue Light Cystoscopy with Cysview after repeated Blue Light Cystoscopy with Cysview evaluations with respect to improved tumor detection, false positive rate and safety compared to conventional white light?
7. Does an abnormal urinalysis help identify patients with inflammation more likely to have false positive Blue Light Cystoscopy with Cysview results?
8. What is the practical learning curve for becoming "proficient" with Blue Light Cystoscopy with Cysview?
9. What is the overall false positive rate with Blue Light Cystoscopy with Cysview?
10. Can Blue Light Cystoscopy with Cysview make the resection more complete? If yes, is this due to improved margins and/or additional tumors seen under blue light?
11. What are the performance characteristics of BLC™ with Cysview® on patients with variant histology?
12. How does BLC™ with Cysview® impact detection of tumors in surveillance and patient management decisions?
13. How does BLC™ with Cysview® impact management of small tumors during office biopsy/fulguration?
14. How can BLC impact patient selection for bladder cancer sparing drugs?
15. Does the combination of BLC with urine biomarkers guide appropriate therapy and or change management?
16. Does BL have an impact on long term outcomes such as recurrence or progression?
17. Can AI models be optimized and validated to accurately predict patient response to intravesical therapy (such as BCG or intravesical chemotherapy) in non-muscle invasive bladder cancer?
18. How concordant are the predictions of AI algorithms with treatment decisions documented in real-world clinical registries?
19. How do AI-predicted responses correlate with patient outcomes, including recurrence and progression, within predefined clinical subgroups such as 'BCG-naïve' or 'no prior intravesical treatment'?
20. What is the potential impact of implementing AI-based predictive models on changes in management (e.g., treatment selection, patient management, and overall care outcomes)?

The Blue Light Cystoscopy with Cysview Registry is a web-based program supported by Global Vision Technologies. Data will be captured longitudinally over five (5) years on patients from each enrolled site. Each center will enter their respective site's patient data electronically.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years old
* Suspected or known non-muscle invasive bladder cancer on the basis of a prior cystoscopy

Exclusion Criteria:

* Porphyria
* Gross hematuria
* Known hypersensitivity to hexaminolevulinate or aminolevulinate derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for transurethral resection of the bladder.
Sampling Method: Probability Sample
Enrollment: 4400 (Estimated)
Dates: Start 2014-04; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of detection of bladder malignancies | 5 years
  Rate of detection of bladder malignancies with Blue Light Cystoscopy with Cysview versus white light cystoscopy alone.

SECONDARY OUTCOMES:
False-positive detection rates | 5 years
  Rates of false-positive lesion biopsies based on pathological findings
Higher-Quality resection rates with Blue Light Cystoscopy with Cysview versus white light cystoscopy alone | 5 years
  Rate of additional margin detection with Blue Light Cystoscopy with Cysview versus white light cystoscopy alone
Proportion of patients with adverse events considered causally related to Cysview in repeat administration. | 5 years
  Adverse events reporting
Recurrence Rates | 5 years
  Recurrence rates NMIBC in patients whose lesions were detected with Blue Light Cystoscopy with Cysview
Cystectomy Rate | 5 years
  Proportion of patients who have a cystectomy performed

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Daneshmand, MD, Principal Investigator — University of Southern California
Locations (23):
- United States (23):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Medicine, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - NYU Langone's Perlmutter Cancer Center, New York, New York
  - Stony Brook Urology, Stony Brook, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Lexington Medical Center, West Columbia, South Carolina
  - UT Southwestern, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - University of Washington Medicine, Seattle, Washington
  - Charleston Area Medical Center, Charleston, West Virginia

REFERENCES:
- [Background] Ghoreifi A, et al. Upstaging and risk migration with blue light cystoscopy for non-muscle-invasive bladder cancer: Results from a prospective multi-center registry. J Clin Oncol. 2025 Feb;43(5 Suppl):686. https://doi.org/10.1200/JCO.2025.43.5_suppl.686
- [Result] Alsyouf M, Ladi-Seyedian SS, Konety B, Pohar K, Holzbeierlein JM, Kates M, Willard B, Taylor JM, Liao JC, Kaimakliotis HZ, Porten SP, Steinberg GD, Tyson MD, Lotan Y, Daneshmand S; Blue Light Cystoscopy with Cysview Registry Group. Is a restaging TURBT necessary in high-risk NMIBC if the initial TURBT was performed with blue light? Urol Oncol. 2023 Feb;41(2):109.e9-109.e14. doi: 10.1016/j.urolonc.2022.10.026. Epub 2022 Nov 24. PMID 36435710
- [Result] Ladi-Seyedian SS, Ghoreifi A, Konety B, Pohar K, Holzbeierlein JM, Taylor J, Kates M, Willard B, Taylor JM, Liao JC, Kaimakliotis HZ, Porten SP, Steinberg GD, Tyson MD, Lotan Y, Daneshmand S, Blue Light Cystoscopy With Cysview Registry Group. Racial Differences in the Detection Rate of Bladder Cancer Using Blue Light Cystoscopy: Insights from a Multicenter Registry. Cancers (Basel). 2024 Mar 24;16(7):1268. doi: 10.3390/cancers16071268. PMID 38610946
- [Result] Perez-Londono A, et al. Performance of the EORTC and CUETO risk prediction models in contemporary patients undergoing transurethral resection of bladder tumor with blue light cystoscopy. J Urol. 2025;213(5 Suppl):e105.
- [Result] Perez-Londono A, et al. Predicting recurrence and progression in contemporary patients with NMIBC undergoing blue light cystoscopy-aided transurethral resection of bladder tumor. J Urol. 2025;213(5 Suppl):e101.
- [Result] Ghoreifi A, Daneshmand S. Technical Considerations to Minimize False-Positive Findings in Blue Light Cystoscopy for Nonmuscle-Invasive Bladder Cancer. J Urol. 2025 Jan;213(1):5-7. doi: 10.1097/JU.0000000000004250. Epub 2024 Sep 16. No abstract available. PMID 39284074
- [Result] Bazargani ST, Shah SH, Djaladat H, et al. Blue Light Cystoscopy For Diagnosis of Urothelial Bladder Cancer: Results: From A Prospective Registry. Poster presented at: The Annual meeting of Society of Urologic Oncology; December 2015; Washington, D.C.
- [Result] Chappidi MR, Yang H, Meng MV, Bivalacqua TJ, Daneshmand S, Holzbeierlein JM, Kaimakliotis HZ, Konety B, Liao JC, Pohar K, Steinberg GD, Taylor JM, Tyson MD, Willard B, Lotan Y, Porten SP, Kates M. Utility of Blue Light Cystoscopy for Post-bacillus Calmette-Guerin Bladder Cancer Recurrence Detection: Implications for Clinical Trial Recruitment and Study Comparisons. J Urol. 2022 Mar;207(3):534-540. doi: 10.1097/JU.0000000000002308. Epub 2021 Oct 25. PMID 34694916
- [Result] Daneshmand S, Patel S, Lotan Y, Pohar K, Trabulsi E, Woods M, Downs T, Huang W, Jones J, O'Donnell M, Bivalacqua T, DeCastro J, Steinberg G, Kamat A, Resnick M, Konety B, Schoenberg M, Jones JS; Flexible Blue Light Study Group Collaborators. Efficacy and Safety of Blue Light Flexible Cystoscopy with Hexaminolevulinate in the Surveillance of Bladder Cancer: A Phase III, Comparative, Multicenter Study. J Urol. 2018 May;199(5):1158-1165. doi: 10.1016/j.juro.2017.11.096. Epub 2017 Dec 2. PMID 29203268
- [Result] Ahmadi H, Ladi-Seyedian SS, Konety B, Pohar K, Holzbeierlein JM, Kates M, Willard B, Taylor JM, Liao JC, Kaimakliotis HZ, Porten SP, Steinberg GD, Tyson MD, Lotan Y, Daneshmand S; Blue Light Cystoscopy with Cysview Registry Group. Role of blue-light cystoscopy in detecting invasive bladder tumours: data from a multi-institutional registry. BJU Int. 2022 Jul;130(1):62-67. doi: 10.1111/bju.15614. Epub 2021 Oct 26. PMID 34637596
- [Result] Daneshmand S, Bazargani ST, Bivalacqua TJ, Holzbeierlein JM, Willard B, Taylor JM, Liao JC, Pohar K, Tierney J, Konety B; Blue Light Cystoscopy with Cysview Registry Group. Blue light cystoscopy for the diagnosis of bladder cancer: Results from the US prospective multicenter registry. Urol Oncol. 2018 Aug;36(8):361.e1-361.e6. doi: 10.1016/j.urolonc.2018.04.013. Epub 2018 May 30. PMID 29859728
- [Result] Matulewicz RS, Ravvaz K, Weissert JA, Porten S, Steinberg GD; Blue Light Cystoscopy with Cysview Registry Group. Association of smoking status and recurrence of non-muscle invasive bladder cancer among patients managed with blue light cystoscopy. Urol Oncol. 2021 Dec;39(12):833.e19-833.e26. doi: 10.1016/j.urolonc.2021.04.028. Epub 2021 May 28. PMID 34053856